CLINICAL TRIAL: NCT02968329
Title: Left Atrial Function as Predictor of Recurrent Stroke or Paroxysmal Atrial Fibrillation in Patients With Cryptogenic Stroke
Brief Title: Left Atrial Function in Recurrent Stroke of Unknown Cause
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, prof. dr., Hasselt University
Other Study IDs: JJBV544
Record Dates: First submitted 2016-11-13; First posted 2016-11-18 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CVA cases: patients who experienced an ischemic CVA or TIA during the study duration and experienced a recurrence.
- CVA controls: patients who experienced an ischemic CVA or TIA during the study duration, but who didn't experience a recurrence.
- AF cases: patients who experienced an ischemic CVA or TIA during the study duration and who got diagnosed with 'new' AF
- AF controls: patients who experienced an ischemic CVA or TIA during the study duration but who didn't get diagnosed with 'new' AF during the study duration

SUMMARY:
Stroke is an important cause of disability and the third leading cause of death.

Approximately 30 to 40 % of all strokes are estimated to be cryptogenic (i.e. no cause can be found). There have been few previous studies regarding risk stratification for stroke recurrence in patients with cryptogenic stroke.

Recent studies have suggested that left atrial (LA) function is an important determinant of stroke risk. However, most studies focus on volume indices and LA dimensions, we also want to investigate other echocardiographic parameters. The aim of this study is to assess the predictive value of left atrial function for the risk of stroke recurrence and/or atrial fibrillation by transthoracic echocardiography in cryptogenic stroke patients with no proven atrial fibrillation (AF) and no indication for anticoagulants.

DETAILED DESCRIPTION:
Study design and population The investigators used a retrospective mono-centric case-control design and analyzed all patients admitted for cerebrovascular accident (CVA) or transient ischemic attack (TIA) between 2011 and 2014. The investigators searched for patients who had a recurrent CVA/TIA and/or who were diagnosed with newly documented AF during the study duration. Clinical, demographic and laboratory parameters were assessed. Echocardiographic parameters, measured on first admission, were analyzed using EchoPAC version 112.

Statistical analysis Univariate analysis was performed for all covariates using the Cox proportional hazards model. Likelihood ratio tests were used to determine significance for all parameters.

If covariates were significant at the 25% significance level, they were used in the multivariate model.

Multivariate analysis was performed using the Cox proportional hazards model with backward elimination model selection. The Wald Chi-Square test was used to determine significance at 5% significance level. The program used for analysis is SAS version 9.4.

ELIGIBILITY:
Inclusion Criteria:

* CVA
* TIA

Exclusion Criteria:

* proven AF or atrial flutter
* prior ablation for AF
* valvular disease
* artificial heart valves
* endocarditis
* presence of an atrial septum defect or moderate to large patent foramen ovale
* LV akinesia
* moderate to severe carotid stenosis
* prior surgery for carotid artery stenosis
* total occlusion of the internal carotid artery
* carotid artery dissection
* vertebral artery dissection
* massive aortic atheromatosis
* temporal arteritis
* basilar artery aneurysm
* ascending aortic aneurysm
* subclavian steal
* prior CVA/TIA
* intracerebral hemorrhage
* lacunar infarction
* clotting disorder
* on anticoagulants
* CVA/TIA as a procedural complication
* hyperthyroidism
* patients who died in hospital after first admission for CVA/TIA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cryptogenic Stroke
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Recurrent ischemic CVA or TIA | up to four years
  Recurrent ischemic CVA or TIA from first ischemic CVA or TIA after 31-12-2010 until date of first documented recurrence, assessed up to four years

SECONDARY OUTCOMES:
'New' diagnosis of AF | Up to four years
  'New' diagnosis of AF from first ischemic CVA or TIA after 31-12-2010 until date of documented 'new' AF, assessed up to four years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dendale, prof. dr., Principal Investigator — Jessa Hospital; Bram Verdonck, student, Study Chair — Hasselt University; Jens Jeurissen, student, Study Chair — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided